CLINICAL TRIAL: NCT05053893
Title: A Randomized, Parallel Controlled Trial of Roxadustat Combined withSacubitril Valsartan Sodium Tablets in the Treatment of Cardiorenal Anemia Syndrome
Brief Title: Roxadustat Combined With Sacubitril Valsartan Sodium Tablets in the Treatment of Cardiorenal Anemia Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Guangqun Xing,MD, Chief physician; Professor, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHASB-001
Record Dates: First submitted 2021-09-12; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Cardio-Renal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — sacubitril and valsartan sodium hydrate drug combination; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New treatment group(Roxadustat combined with Sacubitril Valsartan Sodium Tablets) (Experimental): Roxadustat(FibroGen, China), 100mg (45-60kg) or 120mg (≥ 60kg) each time, three times a week, orally on an empty stomach in the morning. The initial dose of Sacubitril Valsartan Sodium Tablets(Novartis, China) is 50mg, once a day, taken on an empty stomach in the morning, and gradually titrated from the minimum dose to the maximum tolerated dose.
  Interventions: Drug: Roxadustat;Sacubitril Valsartan Sodium Tablets;
- Traditional treatment group(EPO combined with ACEI or ARB ) (Experimental): Recombinant human erythropoietin (SEBOR, 10000 units / Branch) was injected subcutaneously once a week; Perindopril tablets (Servier, China), taken on an empty stomach, gradually titrated from the minimum dose to the maximum tolerated dose.
  Interventions: Drug: EPO; ACEI / ARB

INTERVENTIONS:
Drug: Roxadustat;Sacubitril Valsartan Sodium Tablets; — Select the appropriate dose according to the patient's situation
  Other Names: Entresto®
  Arms: New treatment group(Roxadustat combined with Sacubitril Valsartan Sodium Tablets)
Drug: EPO; ACEI / ARB — Select the appropriate ACEI /ARB according to the subject's situation or follow its previous medication
  Arms: Traditional treatment group(EPO combined with ACEI or ARB )

SUMMARY:
A randomized and parallel controlled trial design of comparing the new treatment group of Roxadustat combined with Sacubitril Valsartan Sodium Tablets with the traditional treatment group of recombinant human erythropoietin (EPO) combined with ACEI or ARB in Chinese patients with cardiorenal anemia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as regular dialysis patients with cardiorenal anemia syndrome
* Hemoglobin 60-110g / L (twice with an interval of at least 4 days);
* Volunteered to participate

Exclusion Criteria:

* Anemia caused by diseases other than CKD
* Malignant tumors
* Active liver disease
* Rheumatic immune diseases in active stage
* Hereditary or idiopathic angioedema
* Systolic blood pressure≥180 mmHg;diastolic blood pressure≥110 mmHg
* Acute myocardial infarction and unstable angina pectoris
* Severe parathyroidism
* Active peptic ulcer
* taking aliskiren
* Mental disease
* Alcohol and drug abuse
* Allergy to test drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-22 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes of hemoglobin level before and after treatment | Day0-Day90
  By detecting blood routine,calculate the changes of hemoglobin.Change value of hemoglobin level(g/L) = baseline hemoglobin level(g/L) - hemoglobin level after treatment(g/L)
Changes of ejection fraction before and after treatment | Day0-Day90
  Cardiac ejection fraction was measured by cardiac ultrasound before and after treatment，and change of cardiac ejection fraction(%) = baseline cardiac ejection fraction level(%) - post-treatment cardiac ejection fraction level(%)
Incidence of acute heart failure, acute myocardial infarction, severe hyperkalemia and severe anemia during treatment | Day0-Day90
  Incidence rate = number of patients with the events/ total number of patients included in the study in this group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Affiliated Hospital of Qingdao University, Qingdao, Shangdong, China